CLINICAL TRIAL: NCT04492657
Title: Study on the Compensatory Mechanism of Iodine Nutrition and the Optimal Intake Level of Lactating Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Wanqi Zhang, professor, Tianjin Medical University
Other Study IDs: NSFC-8191001159
Record Dates: First submitted 2020-07-21; First posted 2020-07-30 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Nutritional Requirements
Keywords: public nutrition; nutrition of special population; lactating women and infants; physiological compensatory mechanism; iodine balance study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood,urine,breast milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — Natural exposure of iodine.

SUMMARY:
Due to the lack of direct evidence of optimal iodine intake of Chinese children, pregnant and lactating women and infants were found during the recent revision of Chinese dietary reference intakes (DRIs) of iodine in 2013 by the applicant Pro. Zhang, and no systematical research about compensatory mechanism of iodine nutrition in lactating women was found yet. Previous study funded by United Nations International Children's Emergency Fund (UNICEF) cooperated with the international experts on iodine and key project of national natural science foundation of China under the guidance of Pro. Zhang, had obtained the safe intake range of iodine from children and pregnant women, more than 10 joint papers were published, which laid the foundation of population study and international cooperation.

DETAILED DESCRIPTION:
Studies indicate lactating women and their infants are the most vulnerable population to the adverse effects of iodine deficiency and excess, and because of the complexity of the study of lactating mothers and infants and the difficulty of sample collection, it is proposed to overcome this problem with the help of the advanced dried blood spot technique and iodine balance study method from the panel of Iodine Global Network (IGN). Investigators intend to recruit 900 late pregnant women in Tianjin, Hebei and Shandong;then establishing a dynamic cohort of breastfeeding mother-infant to 6 months after delivery to investigate the physiological compensatory mechanism of iodine nutrition in lactating women with the combination of animal experiment; On the other hand, 180 exclusively breastfeeding mother and infants within postpartum 0-6 months, will be selected to participate the iodine balance study.

Optimized method of iodine balance experiment of infants by both foreign partner and Pro. Zhang's team will be adopted to obtain the first iodine balance value of Chinese lactating women and infants,providing the direct evidence for the revision of DRIs in lactating women and infants, and guide the lactating women proper iodine supplementation to meet the requirements of both mothers and infants.

ELIGIBILITY:
Inclusion Criteria:

* Women in their third trimester:⑴Aged 18-40, who have lived in the area for 1 year;⑵Single pregnancy;⑶Those who have no special dietary habits;
* Lactating woman:⑴Breastfeeding a child;⑵Normal thyroid function during pregnancy;⑶Term delivery (38-42 weeks of gestation);
* Infants and young children:⑴0-6 months;⑵Breastfeeding;⑶Full term (38-42 weeks of gestation);⑷Normal birth weight (2500-4000g);⑸The thyroid-stimulating hormone (TSH) value of heel blood was normal;⑹Apgar score 8.

Exclusion Criteria:

* Women in their third trimester:⑴Smoking or drinking;⑵Iodized drugs or contrast agents have been used in the past year;⑶A history of thyroid disease, autoimmune disease, endocrine disease, heart disease, chronic disease or family hereditary disease, etc;
* Lactating woman:⑴A history of thyroid disease, autoimmune disease, endocrine disease, heart disease, chronic disease or family hereditary disease, etc;
* Infants and young children:⑴Have pathological jaundice, autoimmune disease, congenital heart disease and other diseases.

Ages: 1 Day to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women in the third trimester (18-40 years old), lactating women (38-42 weeks of gestation) and infants (0-6 months), all from Tianjin, Hebei and Shandong
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Disposable random urine | baseline
  μg/L
Venous blood | baseline
  μg/L
Water iodine intake | baseline
  μg/day
Salt iodine concentration | baseline
  μg/day
Colostrum | 1 week
  μg/L
Mother and child urine randomly at one time | 1 week
  μg/L
Neonatal heel blood | 1 week
  μg/L
Thyroglobulin(TG) | 1 week
  ug/L
Thyroid-stimulating hormone | 1 week
  mIU/L
Infant disposable random urine | 4 weeks
  μg/L
Infant disposable random urine | 24 weeks
  μg/L
Infant disposable random urine | 12 weeks
  μg/L
24 h urine | 4 weeks
  μg/L
24 h urine | 12 weeks
  μg/L
24 h urine | 24 weeks
  μg/L
Urinary iodine excretion | 4 weeks
  μg/day
Urinary iodine excretion | 12 weeks
  μg/day
Urinary iodine excretion | 24 weeks
  μg/day
Milk output | 4 weeks
  μg/day
Milk output | 12 weeks
  μg/day
Milk output | 24 weeks
  μg/day
Milk iodine excretion | 4 weeks
  μg/day
Milk iodine excretion | 12 weeks
  μg/day
Milk iodine excretion | 24 weeks
  μg/day
Average iodine intake | 4 weeks
  μg/day
Average iodine intake | 12 weeks
  μg/day
Average iodine intake | 24 weeks
  μg/day
Thyroid volume | 1 week
  cm³
Thyroid volume | 4 weeks
  cm³
Thyroid volume | 12 weeks
  cm³
Thyroid volume | 24 weeks
  cm³
Thyroid nodule | 1 week
  cm³
Thyroid nodule | 4 weeks
  cm³
Thyroid nodule | 12 weeks
  cm³
Thyroid nodule | 24 weeks
  cm³
Dried blood spot(DBS) | 3 days
  μg/L
Dried blood spot(DBS) | 12 weeks
  μg/L
Diet iodine intake | 1 week
  μg/day
Fecal iodine excretion | 1 week
  μg/day

CONTACTS AND LOCATIONS:
Overall Officials: JianQiang Lai, Principal Investigator — Institute of Nutrition and Health, Chinese Center for Disease Control and Prevention; XueSong Wang, Principal Investigator — Shandong Institute of Endemic Disease Control and Prevention; YiFan Duan, Principal Investigator — Institute of Nutrition and Health, Chinese Center for Disease Control and Prevention; GuiJun Tan, Principal Investigator — Tianjin Medical University; Wen Chen, Principal Investigator — Tianjin Medical University; YanTing Chen, Principal Investigator — Tianjin Medical University; Min Gao, Principal Investigator — Tianjin Medical University; ZiYun Pan, Principal Investigator — Tianjin Medical University; Michael B Zimmermann, doctorate, Study Chair — Swiss federal institute of Technology (ETH); Elizabeth N Pearce, doctorate, Study Chair — Boston University School of Medicine; Iodine Global Network (IGN); Maria Andersson, doctorate, Study Chair — Swiss federal institute of Technology (ETH); Iodine Global Network (IGN)
Locations (4):
- Boston University School of Medicine; Iodine Global Network (IGN), Boston, Massachusetts, United States
- China (2):
  - Institute of Nutrition and Health, Chinese Center for Disease Control and Prevention, Beijing
  - Shandong Institute of Endemic Disease Control and Prevention, Shandong
- Swiss federal institute of Technology (ETH), Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brough L, Thomson BM, Skeaff SA. Revisiting the Iodine Global Network's definition of iodine status by country. Br J Nutr. 2016 Jan 28;115(2):374-6. doi: 10.1017/S0007114515004389. Epub 2015 Dec 2. No abstract available. PMID 26627636
- [Background] Pearce EN, Andersson M, Zimmermann MB. Global iodine nutrition: Where do we stand in 2013? Thyroid. 2013 May;23(5):523-8. doi: 10.1089/thy.2013.0128. Epub 2013 Apr 18. PMID 23472655
- [Background] Sang Z, Wang PP, Yao Z, Shen J, Halfyard B, Tan L, Zhao N, Wu Y, Gao S, Tan J, Liu J, Chen Z, Zhang W. Exploration of the safe upper level of iodine intake in euthyroid Chinese adults: a randomized double-blind trial. Am J Clin Nutr. 2012 Feb;95(2):367-73. doi: 10.3945/ajcn.111.028001. Epub 2011 Dec 28. PMID 22205314
- [Background] Chen W, Li X, Wu Y, Bian J, Shen J, Jiang W, Tan L, Wang X, Wang W, Pearce EN, Zimmermann MB, Carriquiry AL, Zhang W. Associations between iodine intake, thyroid volume, and goiter rate in school-aged Chinese children from areas with high iodine drinking water concentrations. Am J Clin Nutr. 2017 Jan;105(1):228-233. doi: 10.3945/ajcn.116.139725. Epub 2016 Dec 7. PMID 27927635
- [Background] Chen W, Wu Y, Lin L, Tan L, Shen J, Pearce EN, Guo X, Wang W, Bian J, Jiang W, Zhang W. 24-Hour Urine Samples Are More Reproducible Than Spot Urine Samples for Evaluation of Iodine Status in School-Age Children. J Nutr. 2016 Jan;146(1):142-6. doi: 10.3945/jn.115.215806. Epub 2015 Nov 25. PMID 26609173
- [Background] Chen W, Zhang Q, Wu Y, Wang W, Wang X, Pearce EN, Tan L, Shen J, Zhang W. Shift of Reference Values for Thyroid Volume by Ultrasound in 8- to 13-Year-Olds with Sufficient Iodine Intake in China. Thyroid. 2019 Mar;29(3):405-411. doi: 10.1089/thy.2018.0412. PMID 30696370
- [Background] Chen W, Zhang Y, Hao Y, Wang W, Tan L, Bian J, Pearce EN, Zimmermann MB, Shen J, Zhang W. Adverse effects on thyroid of Chinese children exposed to long-term iodine excess: optimal and safe Tolerable Upper Intake Levels of iodine for 7- to 14-y-old children. Am J Clin Nutr. 2018 May 1;107(5):780-788. doi: 10.1093/ajcn/nqy011. PMID 29722836
- [Background] Tan L, Tian X, Wang W, Guo X, Sang Z, Li X, Zhang P, Sun Y, Tang C, Xu Z, Shen J, Zhang W. Exploration of the appropriate recommended nutrient intake of iodine in healthy Chinese women: an iodine balance experiment. Br J Nutr. 2019 Mar 14;121(5):519-528. doi: 10.1017/S0007114518003653. Epub 2018 Dec 11. PMID 30526700
- [Background] Pan Z, Cui T, Chen W, Gao S, Pearce EN, Wang W, Chen Y, Guo W, Tan L, Shen J, Zhang W. Serum iodine concentration in pregnant women and its association with urinary iodine concentration and thyroid function. Clin Endocrinol (Oxf). 2019 May;90(5):711-718. doi: 10.1111/cen.13945. Epub 2019 Mar 7. PMID 30724372
- [Background] Zhang Y, Du C, Wang W, Chen W, Shao P, Wang C, Leng J, Shen J, Tan L, Zhang W. Effect of maternal and neonatal factors on neonatal thyroid stimulating hormone: Results from a population-based prospective cohort study in China. J Trace Elem Med Biol. 2018 Sep;49:151-156. doi: 10.1016/j.jtemb.2018.05.008. Epub 2018 May 25. PMID 29895366
- [Background] Chen Y, Chen W, Du C, Fan L, Wang W, Gao M, Zhang Y, Cui T, Hao Y, Pearce EN, Wang C, Zhang W. Iodine Nutrition and Thyroid Function in Pregnant Women Exposed to Different Iodine Sources. Biol Trace Elem Res. 2019 Jul;190(1):52-59. doi: 10.1007/s12011-018-1530-8. Epub 2018 Oct 2. PMID 30280309
- [Background] Chen W, Sang Z, Tan L, Zhang S, Dong F, Chu Z, Wei W, Zhao N, Zhang G, Yao Z, Shen J, Zhang W. Neonatal thyroid function born to mothers living with long-term excessive iodine intake from drinking water. Clin Endocrinol (Oxf). 2015 Sep;83(3):399-404. doi: 10.1111/cen.12625. Epub 2014 Nov 5. PMID 25280177
- [Background] Sang Z, Wei W, Zhao N, Zhang G, Chen W, Liu H, Shen J, Liu J, Yan Y, Zhang W. Thyroid dysfunction during late gestation is associated with excessive iodine intake in pregnant women. J Clin Endocrinol Metab. 2012 Aug;97(8):E1363-9. doi: 10.1210/jc.2011-3438. Epub 2012 Jun 5. PMID 22669304
- [Background] Stinca S, Andersson M, Herter-Aeberli I, Chabaa L, Cherkaoui M, El Ansari N, Aboussad A, Weibel S, Zimmermann MB. Moderate-to-Severe Iodine Deficiency in the "First 1000 Days" Causes More Thyroid Hypofunction in Infants Than in Pregnant or Lactating Women. J Nutr. 2017 Apr;147(4):589-595. doi: 10.3945/jn.116.244665. Epub 2017 Feb 15. PMID 28202636
- [Background] Bizhanova A, Kopp P. Minireview: The sodium-iodide symporter NIS and pendrin in iodide homeostasis of the thyroid. Endocrinology. 2009 Mar;150(3):1084-90. doi: 10.1210/en.2008-1437. Epub 2009 Feb 5. PMID 19196800
- [Background] Suzuki K, Kimura H, Wu H, Kudo N, Kim WB, Suzuki S, Yoshida A, Caturegli P, Kohn LD. Excess iodide decreases transcription of NIS and VEGF genes in rat FRTL-5 thyroid cells. Biochem Biophys Res Commun. 2010 Mar 5;393(2):286-90. doi: 10.1016/j.bbrc.2010.01.123. Epub 2010 Feb 2. PMID 20132794
- [Background] Dold S, Zimmermann MB, Baumgartner J, Davaz T, Galetti V, Braegger C, Andersson M. A dose-response crossover iodine balance study to determine iodine requirements in early infancy. Am J Clin Nutr. 2016 Sep;104(3):620-8. doi: 10.3945/ajcn.116.134049. Epub 2016 Jul 27. PMID 27465383
- [Background] Kleinau G, Biebermann H. Constitutive activities in the thyrotropin receptor: regulation and significance. Adv Pharmacol. 2014;70:81-119. doi: 10.1016/B978-0-12-417197-8.00003-1. PMID 24931193
- [Background] Van Sande J, Dequanter D, Lothaire P, Massart C, Dumont JE, Erneux C. Thyrotropin stimulates the generation of inositol 1,4,5-trisphosphate in human thyroid cells. J Clin Endocrinol Metab. 2006 Mar;91(3):1099-107. doi: 10.1210/jc.2005-1324. Epub 2005 Dec 29. PMID 16384841
- [Background] Thomasz L, Oglio R, Salvarredi L, Perona M, Rossich L, Copelli S, Pisarev M, Juvenal G. Regulation of NADPH oxidase NOX4 by delta iodolactone (IL-delta) in thyroid cancer cells. Mol Cell Endocrinol. 2018 Jul 15;470:115-126. doi: 10.1016/j.mce.2017.10.004. Epub 2017 Oct 7. PMID 28993239
- [Background] Calil-Silveira J, Serrano-Nascimento C, Kopp PA, Nunes MT. Iodide excess regulates its own efflux: a possible involvement of pendrin. Am J Physiol Cell Physiol. 2016 Apr 1;310(7):C576-82. doi: 10.1152/ajpcell.00210.2015. Epub 2016 Jan 20. PMID 26791486
- [Background] Perron B, Rodriguez AM, Leblanc G, Pourcher T. Cloning of the mouse sodium iodide symporter and its expression in the mammary gland and other tissues. J Endocrinol. 2001 Jul;170(1):185-96. doi: 10.1677/joe.0.1700185. PMID 11431151
- [Background] Ryan J, Curran CE, Hennessy E, Newell J, Morris JC, Kerin MJ, Dwyer RM. The sodium iodide symporter (NIS) and potential regulators in normal, benign and malignant human breast tissue. PLoS One. 2011 Jan 19;6(1):e16023. doi: 10.1371/journal.pone.0016023. PMID 21283523
- [Background] Nicola JP, Reyna-Neyra A, Carrasco N, Masini-Repiso AM. Dietary iodide controls its own absorption through post-transcriptional regulation of the intestinal Na+/I- symporter. J Physiol. 2012 Dec 1;590(23):6013-26. doi: 10.1113/jphysiol.2012.241307. Epub 2012 Sep 24. PMID 23006481
- [Background] De la Vieja A, Santisteban P. Role of iodide metabolism in physiology and cancer. Endocr Relat Cancer. 2018 Apr;25(4):R225-R245. doi: 10.1530/ERC-17-0515. Epub 2018 Feb 1. PMID 29437784
- [Background] Yu X, Shen H, Liu L, Lin L, Gao M, Wang S. Changes of sodium iodide symporter regulated by IGF-I and TGF-beta1 in mammary gland cells from lactating mice at different iodine levels. Biol Trace Elem Res. 2012 Apr;146(1):73-8. doi: 10.1007/s12011-011-9227-2. Epub 2011 Oct 13. PMID 21993965
- [Background] Huynh D, Condo D, Gibson R, Muhlhausler B, Ryan P, Skeaff S, Makrides M, Zhou SJ. Iodine status of postpartum women and their infants in Australia after the introduction of mandatory iodine fortification. Br J Nutr. 2017 Jun;117(12):1656-1662. doi: 10.1017/S0007114517001775. PMID 28789730
- [Background] Chung HR, Shin CH, Yang SW, Choi CW, Kim BI. Subclinical hypothyroidism in Korean preterm infants associated with high levels of iodine in breast milk. J Clin Endocrinol Metab. 2009 Nov;94(11):4444-7. doi: 10.1210/jc.2009-0632. Epub 2009 Oct 6. PMID 19808851
- [Background] Liu L, Wang D, Liu P, Meng F, Wen D, Jia Q, Liu J, Zhang X, Jiang P, Shen H. The relationship between iodine nutrition and thyroid disease in lactating women with different iodine intakes. Br J Nutr. 2015 Nov 14;114(9):1487-95. doi: 10.1017/S0007114515003128. Epub 2015 Sep 14. PMID 26365041
- [Background] Aakre I, Bjoro T, Norheim I, Strand TA, Barikmo I, Henjum S. Excessive iodine intake and thyroid dysfunction among lactating Saharawi women. J Trace Elem Med Biol. 2015;31:279-84. doi: 10.1016/j.jtemb.2014.09.009. Epub 2014 Oct 6. PMID 25447589
- [Background] Nazeri P, Zarghani NH, Mirmiran P, Hedayati M, Mehrabi Y, Azizi F. Iodine Status in Pregnant Women, Lactating Mothers, and Newborns in an Area with More Than Two Decades of Successful Iodine Nutrition. Biol Trace Elem Res. 2016 Jul;172(1):79-85. doi: 10.1007/s12011-015-0575-1. Epub 2015 Dec 2. PMID 26631051
- [Background] Dold S, Zimmermann MB, Aboussad A, Cherkaoui M, Jia Q, Jukic T, Kusic Z, Quirino A, Sang Z, San Luis TO, Vandea E, Andersson M. Breast Milk Iodine Concentration Is a More Accurate Biomarker of Iodine Status Than Urinary Iodine Concentration in Exclusively Breastfeeding Women. J Nutr. 2017 Apr;147(4):528-537. doi: 10.3945/jn.116.242560. Epub 2017 Feb 22. PMID 28228508
- [Background] Nazeri P, Dalili H, Mehrabi Y, Hedayati M, Mirmiran P, Azizi F. Breast Milk Iodine Concentration Rather than Maternal Urinary Iodine Is a Reliable Indicator for Monitoring Iodine Status of Breastfed Neonates. Biol Trace Elem Res. 2018 Sep;185(1):71-77. doi: 10.1007/s12011-018-1246-9. Epub 2018 Jan 25. PMID 29372437
- [Background] Henjum S, Kjellevold M, Ulak M, Chandyo RK, Shrestha PS, Froyland L, Strydom EE, Dhansay MA, Strand TA. Iodine Concentration in Breastmilk and Urine among Lactating Women of Bhaktapur, Nepal. Nutrients. 2016 Apr 28;8(5):255. doi: 10.3390/nu8050255. PMID 27136582
- [Background] Chan SS, Hams G, Wiley V, Wilcken B, McElduff A. Postpartum maternal iodine status and the relationship to neonatal thyroid function. Thyroid. 2003 Sep;13(9):873-6. doi: 10.1089/105072503322401078. PMID 14588102
- [Background] Wang W, Sun Y, Zhang M, Zhang Y, Chen W, Tan L, Shen J, Zhao Z, Lan S, Zhang W. Breast milk and infant iodine status during the first 12 weeks of lactation in Tianjin City, China. Asia Pac J Clin Nutr. 2018;27(2):393-398. doi: 10.6133/apjcn.062017.03. PMID 29384328
- [Background] Henjum S, Barikmo I, Strand TA, Oshaug A, Torheim LE. Iodine-induced goitre and high prevalence of anaemia among Saharawi refugee women. Public Health Nutr. 2012 Aug;15(8):1512-8. doi: 10.1017/S1368980011002886. Epub 2011 Nov 7. PMID 22053869
- [Background] Dworkin HJ, Jacquez JA, Beierwaltes WH. Relationship of iodine ingestion to iodine excretion in pregnancy. J Clin Endocrinol Metab. 1966 Dec;26(12):1329-42. doi: 10.1210/jcem-26-12-1329. No abstract available. PMID 5959526
- [Background] Institute of Medicine (US) Panel on Micronutrients. Dietary Reference Intakes for Vitamin A, Vitamin K, Arsenic, Boron, Chromium, Copper, Iodine, Iron, Manganese, Molybdenum, Nickel, Silicon, Vanadium, and Zinc. Washington (DC): National Academies Press (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK222310/ PMID 25057538
- [Background] Zimmermann MB, de Benoist B, Corigliano S, Jooste PL, Molinari L, Moosa K, Pretell EA, Al-Dallal ZS, Wei Y, Zu-Pei C, Torresani T. Assessment of iodine status using dried blood spot thyroglobulin: development of reference material and establishment of an international reference range in iodine-sufficient children. J Clin Endocrinol Metab. 2006 Dec;91(12):4881-7. doi: 10.1210/jc.2006-1370. Epub 2006 Sep 12. PMID 16968789
- [Background] Zimmermann MB, Moretti D, Chaouki N, Torresani T. Development of a dried whole-blood spot thyroglobulin assay and its evaluation as an indicator of thyroid status in goitrous children receiving iodized salt. Am J Clin Nutr. 2003 Jun;77(6):1453-8. doi: 10.1093/ajcn/77.6.1453. PMID 12791623
- [Background] Farebrother J, Zimmermann MB, Assey V, Castro MC, Cherkaoui M, Fingerhut R, Jia Q, Jukic T, Makokha A, San Luis TO, Wegmuller R, Andersson M. Thyroglobulin Is Markedly Elevated in 6- to 24-Month-Old Infants at Both Low and High Iodine Intakes and Suggests a Narrow Optimal Iodine Intake Range. Thyroid. 2019 Feb;29(2):268-277. doi: 10.1089/thy.2018.0321. PMID 30648484
- [Background] Ingenbleek Y, Malvaux P. Iodine balance studies in protein-calorie malnutrition. Arch Dis Child. 1974 Apr;49(4):305-9. doi: 10.1136/adc.49.4.305. PMID 4208456
- [Background] Knudsen N, Bulow I, Jorgensen T, Perrild H, Ovesen L, Laurberg P. Serum Tg--a sensitive marker of thyroid abnormalities and iodine deficiency in epidemiological studies. J Clin Endocrinol Metab. 2001 Aug;86(8):3599-603. doi: 10.1210/jcem.86.8.7772. PMID 11502784
- [Background] Zimmermann MB, Aeberli I, Andersson M, Assey V, Yorg JA, Jooste P, Jukic T, Kartono D, Kusic Z, Pretell E, San Luis TO Jr, Untoro J, Timmer A. Thyroglobulin is a sensitive measure of both deficient and excess iodine intakes in children and indicates no adverse effects on thyroid function in the UIC range of 100-299 mug/L: a UNICEF/ICCIDD study group report. J Clin Endocrinol Metab. 2013 Mar;98(3):1271-80. doi: 10.1210/jc.2012-3952. Epub 2013 Jan 23. PMID 23345097
- [Background] Yan YQ, Dong ZL, Dong L, Wang FR, Yang XM, Jin XY, Lin LX, Sun YN, Chen ZP. Trimester- and method-specific reference intervals for thyroid tests in pregnant Chinese women: methodology, euthyroid definition and iodine status can influence the setting of reference intervals. Clin Endocrinol (Oxf). 2011 Feb;74(2):262-9. doi: 10.1111/j.1365-2265.2010.03910.x. PMID 21044115
- [Background] Mao IF, Ko YC, Chen ML. The stability of iodine in human sweat. Jpn J Physiol. 1990;40(5):693-700. doi: 10.2170/jjphysiol.40.693. PMID 2086989
- [Background] Swanson CA, Zimmermann MB, Skeaff S, Pearce EN, Dwyer JT, Trumbo PR, Zehaluk C, Andrews KW, Carriquiry A, Caldwell KL, Egan SK, Long SE, Bailey RL, Sullivan KM, Holden JM, Betz JM, Phinney KW, Brooks SP, Johnson CL, Haggans CJ. Summary of an NIH workshop to identify research needs to improve the monitoring of iodine status in the United States and to inform the DRI. J Nutr. 2012 Jun;142(6):1175S-85S. doi: 10.3945/jn.111.156448. Epub 2012 May 2. PMID 22551802
- [Derived] Zhang Y, Zhao X, Meng H, Jia X, Zhang Z, Zuo Z, He X, Wu P, Jiang X, Zhang W, Sang Z. Estimation of iodine nutrition status among lactating women with adequate iodine based on fractional iodine excretion in urine. Br J Nutr. 2025 Aug 28;134(4):297-303. doi: 10.1017/S0007114525104170. Epub 2025 Aug 12. PMID 40790513
- [Derived] Li S, Wang C, Cheng Y, Li J, Zhang H, Jin Q, Meng Q, Wu W, Wang T, Liu D, Meng X, Guo W, Zhang W. Iodine Metabolism in Urine and Breast Milk among Lactating Women with Adequate Iodine. J Nutr. 2024 Jul;154(7):2006-2013. doi: 10.1016/j.tjnut.2024.04.041. Epub 2024 May 6. PMID 38718924
- [Derived] Li S, Guo W, Jin Q, Meng Q, Yang R, Zhang H, Fu M, Wang T, Liu D, Meng X, Zhang W. Salivary iodine concentration in pregnant women and its association with iodine status and thyroid function. Eur J Nutr. 2024 Jun;63(4):1139-1149. doi: 10.1007/s00394-024-03332-y. Epub 2024 Feb 14. PMID 38355932